CLINICAL TRIAL: NCT03399266
Title: Mechanical Induction of Labor in Women With Previous Cesarean Section and Premature Rupture of Membranes Who Desire TOLAC: A Prospective Randomized Study
Brief Title: Balloon Induction of Labor in PROM for TOLAC
Acronym: BILROM-TOLAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Gil Gutvirtz MD, Ob/Gyn Resident, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR-0019-17-CTIL
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Previous; Cesarean Section, Cicatricial, Complicating Pregnancy or Childbirth, Affecting Fetus or Newborn; Prelabor Rupture of Membranes
Keywords: Induction of labor; Previous cesarean delivery; Trial of labor after cesarean; Prelabor rupture of membranes; balloon induction
MeSH Terms: conditions — Pregnancy Complications; Fetal Membranes, Premature Rupture | interventions — Labor, Induced

STUDY DESIGN:
Intervention Model Description: 200 pregnant women with one previous cesarean section and PROM along with an unfavourable cervix (Bishop Score ≤ 6) are expected to be entered into the study.
  All eligible women will be presented with the study protocol by a study coordinator.The following screening medical procedures will be completed:
  Medical and gynecological history, physical and vaginal speculum examination, Ultrasonography and a non-stress test (NST).
  For eligible patients, and following an informed consent, group randomization will take place:
  GROUP 1: Expectant management (standard protocol). GROUP 2: Insertion of a balloon cervical catheter (study group).
  The randomization process will be as follows:
  A. The eligible patient will sign the informed consent prior to randomization. B. The patient will receive a subject number for the study (from 1 to 200) The study coordinator will open a sealed envelope with the patient's study number to reveal the patient's assigned study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double balloon catheter for induction of labor (Experimental): in this group a trans-cervical double balloon catheter will be inserted. Following device insertion, 20 minutes of external monitoring is performed. The patient will be transferred to the Ob/Gyn ward for hospitalization. 12 hours after insertion of the device the balloons are deflated and the device removed. At this stage the patient is assessed for a second Bishop score and expectant management is resuming.
  Interventions: Device: Double Balloon catheter for induction of labor
- Expectant management (No Intervention): Women in the expectant management group will be transferred to the Ob/Gyn ward for hospitalization and conservative management until spontaneous labor ensues.

INTERVENTIONS:
Device: Double Balloon catheter for induction of labor — With the patient in lithotomy position or lying supine in bed, a speculum is inserted to visualise the cervix. The device is inserted into the cervix using long forceps until both balloons enter the cervical canal. Then, the uterine balloon is inflated with 20 ml of saline (by means of a 20 ml syringe). The device is then pulled out until stopped by the uterine balloon covering the internal cervical os. At this point the cervico-vaginal balloon located at the external os is inflated with 20 ml of saline and the speculum is removed. Then both balloons are additionally inflated with alternate increments of 20 ml normal saline to a total volume of 80 ml in each balloon. The device is loosely taped to the patient's inner thigh.
  Other Names: Atad Ripener Device
  Arms: Double balloon catheter for induction of labor

SUMMARY:
A prospective randomized controlled trial to evaluate the safety and efficacy of labor induction with a double balloon catheter (Atad Ripener Device) in women desiring TOLAC (trial of labor after cesarean) with PROM (pre labor rupture of membranes).

ELIGIBILITY:
Inclusion Criteria:

Only patients who meet the following criteria will be approached.

1. Singleton Pregnancy
2. Previous single cesarean section
3. At least 12 months have elapsed since the previous caesarean delivery
4. Diagnosed with confirmed PROM at ≥ 34 weeks' gestation.
5. Ruptured membranes have occurred ≤24 hours prior to inclusion in the study.
6. Vertex presentation well applied to the cervix
7. Found to have an unripe cervix in a speculum examination (Bishop score ≤6).
8. Absence of significant and regular uterine contraction (<3/10Min).
9. Willingness to comply with the protocol for the duration of the study.
10. Have signed an informed consent (including a TOLAC consent form).

Exclusion Criteria:

Patients having any of the following conditions will be excluded from the study:

1. Any contraindication for a vaginal delivery (i.e. placenta previa, non-vertex presentation, previous cesarean delivery < 12 months).
2. Regular uterine contractions (>3/10Min).
3. Diagnosis of ruptured membranes was made over 24 hours prior to study inclusion.
4. Meconium stained amniotic fluid.
5. Evidence of chorio-amnionitis (T 37.6°C with uterine tenderness and maternal or fetal tachycardia or purulent discharge or WBC20.000)
6. Suspected placental abruption or a significant hemorrhage.
7. Non-reassuring fetal status (as determined by fetal heart rate monitoring and/or bio-physical profile) necessitating immediate intervention.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Vaginal birth after cesarean (VBAC) rates | 5 days

SECONDARY OUTCOMES:
PROM to delivery interval (time) | 5 days
intrapartum and post-partum infection rates | 5 days
Cesarean section rates | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264